CLINICAL TRIAL: NCT00893308
Title: Metabolic Viral Host Properties
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Yaron Ilan, Hadassah medical organization
Other Study IDs: 481133- HMO-CTIL
Record Dates: First submitted 2009-04-26; First posted 2009-05-06 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Patients' metabolic properties may affect their immune response. This study aims to assess the effect of hosts' metabolic properties to viral infection.

DETAILED DESCRIPTION:
Blood samples were drawn from patients with Gaucher disease and healthy individuals, with and without HCV. Blood samples were tested for protein specific T cell proliferation, IFNg and IL-10 using ELISPOT assays, serum IFNg, IL-2, IL-6, IL-10 and IL-4 levels. FACS analysis was used for evaluation of lymphocytes subsets.

ELIGIBILITY:
Inclusion Criteria:

* inform consent

Exclusion Criteria:

* at patients request

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both male and female volunteers were recruited. with and without HCV infection, with and without Gaucher disease.
Sampling Method: Non-Probability Sample